CLINICAL TRIAL: NCT00762476
Title: A MULTI-CENTER, DOUBLE-BLIND, PLACEBO-CONTROLLED PHASE II EFFICACY TRIAL OF AV LOTION (FORMULA NO. 3804-250A) FOR THE PREVENTION OF COLD ILLNESS IN HUMAN SUBJECTS
Brief Title: Efficacy Trial of 3804-250A in the Prevention of Cold Illnesses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Dial Corporation (Industry)
Collaborators: Hill Top Research (Industry); TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TM&R-0062-08-TXC; CS990108; 13805
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-03

CONDITIONS: Common Cold
Keywords: cold, common; rhinovirus
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: 3804-291
- 3804-250A (Experimental)
  Interventions: Drug: 3804-250A

INTERVENTIONS:
Drug: 3804-250A — * topical product
  * apply 2 pumps
  * apply at least every 4 hours or after hand washing
  Arms: 3804-250A
Drug: 3804-291 — * topical
  * apply 2 pumps
  * apply at least every 4 hours or after hand washing
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of 3804-250A in the prevention of the common cold. The study will also evaluate whether 3804-250A prevents rhinovirus infection, a virus that causes many common colds.

DETAILED DESCRIPTION:
Rhinovirus infections are the most frequent cause up to 80% of cold illnesses during the fall rhinovirus season. While viral upper respiratory infections are generally mild and self-limited, they are associated with an enormous economic burden both in lost productivity and in expenditures for treatment. Rhinovirus infection is frequently associated with medical complications that have substantial morbidity such as acute otitis media and exacerbation of asthma.

Marketed treatment options for rhinovirus consist primarily of symptomatic cold remedies have only modest effects on specific cold symptoms. 3804-250A is under investigation for the prevention of rhinovirus infection by interruption of person-to-person transmission appears to be technologically and economically feasible.

The study is a randomized, double-blind, Placebo controlled, multi-site, parallel design clinical trial conducted in the natural setting. The study will be conducted during a 10-week period during the fall rhinovirus epidemic season. Healthy, normal subjects will be recruited and randomly assigned to the AV Lotion or Placebo control group. Subjects will use the assigned test product on a defined schedule and will record the presence of cold illness symptoms daily. Subjects will return to the study site every week during the study for review and clarification of study diary entries, for review and assessment of compliance, for specimen collection for rhinovirus PCR.

ELIGIBILITY:
Inclusion Criteria:

* healthy normal
* good general health

Exclusion Criteria:

* pregnancy
* insulin dependent diabetes
* daily smoker
* skin disease on the hands/wrists
* immunological disorders
* occupation involving frequent handwashing
* common cold symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Turner, MD, Principal Investigator — University of Virginia School of Medicine; Michael E Casser, MD, Principal Investigator — TKL Research, Inc.
Locations (2):
- United States (2):
  - TKL Research, Inc., Paramus, New Jersey
  - University of Virginia School of Medicine, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Modified AV Lotion without active ingredients.
- 3804-250A: Experimental AV Lotion
Period: Overall Study
Arm/Group | Placebo | 3804-250A
Started | 206 | 205
Completed | 183 | 169
Not Completed | 23 | 36
Not completed — Adverse Event | 7 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 5 | 6
Not completed — Physician Decision | 2 | 14
Not completed — Withdrawal by Subject | 6 | 12
Not completed — antibiotic use | 0 | 1
Not completed — non-compliance with study visits | 0 | 2
Not completed — Seasonal allergies | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 3804-250A | Total
Number analyzed (Participants) | 206 | 205 | 411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 203 | 200 | 403
  >=65 years | 3 | 5 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (14.56) | 36.2 (14.23) | 36.7 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 155 | 305
  Male | 56 | 50 | 106
Region of Enrollment [Number; unit: participants]
  United States | 206 | 205 | 411

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint of This Study is the Incidence of Cold Illnesses.
Description: Comparison of the total number of incidence of cold illnesses over the course of the study per 100 subjects in each treatment group
Time Frame: 10 weeks
Population: All efficacy analyses were performed on the intent-to-treat (ITT).The ITT population included all enrolled subjects who received study treatment.
Measure: Number; unit: cold illnesses per 100 subjects
Arm/Group | Placebo | 3804-250A
Number analyzed (Participants) | 206 | 205
cold illnesses per 100 subjects | 47.1 | 43.9
Statistical Analysis 1: Comparison: Placebo vs 3804-250A; Test type: Superiority or Other; p > 0.5000, Poisson regression

2. Secondary Outcome: Rhinovirus Infections.
Description: The incidence of rhinovirus infections
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: rhinovirus infections per 100 subjects
Arm/Group | Placebo | 3804-250A
Number analyzed (Participants) | 206 | 205
rhinovirus infections per 100 subjects | 58.7 | 59.0
Statistical Analysis 1: Comparison: Placebo vs 3804-250A; Test type: Superiority or Other; p > 0.5000, Poisson regression

3. Secondary Outcome: Rhinovirus-associated Colds
Description: The incidence of rhinovirus-associated cold illnesses.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: RV-associated cold illnesses per 100 sub
Arm/Group | Placebo | 3804-250A
Number analyzed (Participants) | 206 | 205
RV-associated cold illnesses per 100 sub | 24.3 | 20.0
Statistical Analysis 1: Comparison: Placebo vs 3804-250A; Test type: Superiority or Other; p = 0.3451, Poisson regression

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo | 3804-250A
Serious Adverse Events (participants affected / at risk) | 2/206 | 0/205
Other Adverse Events (participants affected / at risk) | 23/206 | 16/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=206) | 3804-250A (N=205)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Injury secondary to motor vehicle accident
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) — Injury secondary to motor vehicle accident
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Affected C1 & C3 vertebra. Injury secondary to motor vehicle accident.
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Left side of neck and head affected. Injury secondary to motor vehicle accident.
excoriation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) — Left forehead and left cheek affected. Injury secondary to motor vehicle accident.
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=206) | 3804-250A (N=205)
Application site pruritus (General disorders) | 1 (2) | 7 (8)
Application site vesicles (General disorders) | 2 (2) | 4 (6)
Skin laceration (Injury, poisoning and procedural complications) | 23 (32) | 16 (20)
Excoriation (Injury, poisoning and procedural complications) | 14 (22) | 13 (21)
thermal burn (Injury, poisoning and procedural complications) | 12 (13) | 8 (9)
Scratch (Injury, poisoning and procedural complications) | 7 (8) | 7 (9)
Open wound (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 8 (11) | 6 (7)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (7) | 1 (1)
Oral herpes (Infections and infestations) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period 1 year after study completion.